CLINICAL TRIAL: NCT01304173
Title: A Retrospective Analysis to Evaluate the Effectiveness, Safety and Tolerability of Intravesical Valrubicin for the Treatment of Bladder Carcinoma in Situ in Clinical Practice
Brief Title: Retrospective Chart Review of Valstar
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3329-401
Record Dates: First submitted 2011-02-23; First posted 2011-02-25 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Carcinoma in Situ of Bladder
Keywords: BCG; refractory; NMIBC; CIS; non-muscle invasive
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study involving a retrospective review of medical records of adult patients who have been treated with intravesical valrubicin for bladder carcinoma in situ (CIS) since October 2009.

DETAILED DESCRIPTION:
Initial treatment for bladder CIS is TURBT followed by intravesical immunotherapy with BCG. Valrubicin is approved by the FDA for the treatment of BCG-refractory bladder CIS in patients for whom immediate cystectomy would be associated with unacceptable morbidity or mortality. The recommended course of therapy is 6 doses of 800 mg each administered intravesically once a week. While the benefit risk profile of valrubicin has been established in several clinical trials, current data on effectiveness and tolerability when used in clinical practice are lacking. This protocol outlines a retrospective study to evaluate the effectiveness, safety and tolerability of intravesical valrubicin in the treatment of NMIBC in a clinical practice setting.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or greater
* diagnosis of CIS (physician defined in the medical record)
* treated with at least one IVe dose of valrubicin since 10/2009 and completed prescribed therapy or no longer receiving therapy at time of study enrollment
* willing and able to provide informed consent (unless waiver of informed consent is applicable and in place at that clinical site per Chapter 45 CFR part 46 Subpart A 46.117

Exclusion Criteria:

* route of administration of valrubicin other than intravesical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with valrubicin in a clinical practice setting.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Event-free survival | 12 months
  Event-free survival defined as recurrence, progression or death from any cause

SECONDARY OUTCOMES:
Worsening-free Survival | 12 months
  Worsening-free survival defined as recurrence, progression, cystectomy, change of anti-bladder cancer therapy or death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cookson, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States